CLINICAL TRIAL: NCT06310174
Title: A Pilot Study Examining the Effect of a Novel Cannulation Knife on User Satisfaction and Common Central Venous Catheter Insertion Complications
Brief Title: Study Examining the Effect of a Novel Cannulation Knife on User Satisfaction and Common Central Venous Catheter Insertion Complications
Acronym: SCAD
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00362883
Record Dates: First submitted 2024-03-07; First posted 2024-03-15 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Central Venous Catheter Exit Site Infection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to assess user satisfaction and the frequency of common central venous catheter insertion complications when using a novel cannulation knife.

DETAILED DESCRIPTION:
The primary objective is to assess user satisfaction with a new cannulation knife for central venous catheter (CVC) insertion. Secondary objectives include assessing the frequency of skin incision revisions, frequency of procedures being aborted and restarted, frequency of reverting to the use of the scalpel customarily used to make the incision, frequency of bleeding around the catheter after completion of the procedure, assessment of time to final catheter placement, and the frequency of central line-associated bloodstream infections (CLABSI).

The cannulation knife will be studied in three clinical areas:

* Cardiovascular Operating Room
* Cardiovascular Surgical Intensive Care Unit
* Interventional Cardiology

A prospective cohort of 24 clinicians will be enrolled. Each clinician will be asked to perform a total of five observed cannulations, resulting in a combined 120 observed procedures.

In cases where both the clinician and patient are amenable, a video recording will be taken of the procedure to document the study variables of interest (duration of the procedure, need for revisions, the incidence of bleeding, size of the final incision, etc.) and allow for later review.

All clinicians will be given a survey. This survey is designed to assess the clinicians impression of the device's benefit and the need for 1) revisions of the incision or, 2) aborting the initial attempt. Clinicians will also be timed from procedure start to final catheter placement and will be monitored for incidence of common complications (back bleeding around the catheter, need to revise incision, need to abort/restart procedure) and need to revert to use of a standard scalpel. Although clinicians are the primary focus of this investigation, patients will also be consented to the study and will be monitored for the development of CLABSI post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patient requires a 5 French, 7 French, or 12-14 French central venous catheter.
* Operator responsible for insertion of central venous catheter.

Exclusion Criteria:

* Patient unwilling to consent.
* Operator unwilling to complete the survey.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A prospective cohort of 100 clinicians will be enrolled.
  The cannulation knife will be studied in three clinical areas:
  * Cardiovascular Operating Room
  * Cardiovascular Surgical Intensive Care Unit
  * Interventional Cardiology
Sampling Method: Non-Probability Sample
Enrollment: 144 (Estimated)
Dates: Start 2023-12-22 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
User satisfaction with the new cannulation knife for CVC insertion. | Within one (1) hour post-procedure
  Using a survey developed by the study team, Operators will rate the performance of the cannulation knife in regards to the ease of skin incision, ease of dilator insertion, device safety, and opinion on usage for central venous line (CVL) placement with ongoing cardiopulmonary resuscitation (CPR), using a Likert Scale (scores range from 1: significant benefit to 5: significant hindrance). The possible overall score ranges from four (4) to twenty (20), with a higher score indicating user dissatisfaction and hindrance.

SECONDARY OUTCOMES:
Frequency of skin incision revisions. | Within one (1) hour post-procedure
  Operator will answer: Did you have to revise the incision? Yes No
Frequency of procedures being aborted and restarted. | Within one (1) hour post-procedure
  Operator will answer: Did you have to abort the procedure and start over? Yes No
Frequency of reverting to use of the scalpel normally used to make the incision. | Within one (1) hour post-procedure
  Did you have to revert to using an #11 blade?
Presence of a clean, dry dressing. | Within thirty-six hours (36) post-procedure
  Is dressing dry, clean, and intact?

CONTACTS AND LOCATIONS:
Overall Officials: James Gammie, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States